CLINICAL TRIAL: NCT07012343
Title: Exploring Different Dose-frequency Home Photodynamic Therapy Protocols Using a Novel Home-targeted LED Device for Onychomycosis, a Randomized Feasibility Trial.
Brief Title: Exploring Different Dose-frequency Home Photodynamic Therapy Protocols Using a Novel Home-targeted LED Device for Onychomycosis
Acronym: HomePDT_Nails
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Health Systems Research Institute,Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CUHomePhod_Onychomycosis
Record Dates: First submitted 2025-05-31; First posted 2025-06-10 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-05

CONDITIONS: Onychomycosis of Toenails; Onychomycosis of Fingernail
Keywords: Onychomycosis; Photodynamic therapy; Methylene blue; home phototherapy; portable device
MeSH Terms: conditions — Onychomycosis | interventions — Photochemotherapy; Urea

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- PDT_160OIW (Experimental): once a week of MB-PDT at 160/cm2 and 40%Urea cream with occlusion before MB-PDT
  Interventions: Radiation: Photodynamic Therapy with Conventional Methylene Blue; Drug: urea 40% cream
- PDT_160BIW (Experimental): Twice a week of MB-PDT at 160/cm2 and 40%Urea cream with occlusion before MB-PDT
  Interventions: Radiation: Photodynamic Therapy with Conventional Methylene Blue; Drug: urea 40% cream
- PDT_120BIW (Experimental): Twice a week of MB-PDT at 120/cm2 and 40%Urea cream with occlusion before MB-PDT
  Interventions: Radiation: Photodynamic Therapy with Conventional Methylene Blue; Drug: urea 40% cream
- PDT_80BIW (Experimental): Twice a week of MB-PDT at 80/cm2 and 40%Urea cream with occlusion before MB-PDT
  Interventions: Radiation: Photodynamic Therapy with Conventional Methylene Blue; Drug: urea 40% cream
- NonPDT (Placebo Comparator): 40%Urea cream with occlusion
  Interventions: Drug: urea 40% cream

INTERVENTIONS:
Radiation: Photodynamic Therapy with Conventional Methylene Blue — Methylene Blue mediated photodynamic therapy
  Arms: PDT_120BIW; PDT_160BIW; PDT_160OIW; PDT_80BIW
Drug: urea 40% cream — 40% Urea cream with occlusion

SUMMARY:
This randomized feasibility trial aims to determine the optimal light energy dose and treatment frequency for home-based photodynamic therapy (hPDT) using a novel LED device (L-Home PhoD) for the treatment of onychomycosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with onychomycosis (nail fungal infection) by a dermatologist.
* Diagnosis criteria include at least one clinical criterion combined with at least one laboratory examination criterion.

Clinical Criteria:

* Discoloration patches/streaks on the nail.
* Onycholysis (nail separation from the nail bed).
* Subungual hyperkeratosis/debris (thickening under the nail).
* Nail plate thickening.
* Laboratory Examination Criteria:
* Direct microscopy using KOH preparation.
* Histopathological examination using Periodic Acid Schiff (PAS) stain.
* Patients with distal lateral subungual onychomycosis (DLSO) of the fingernails or toenails, except for the little toenail.
* Patients with onychomycosis who have limitations on or refuse oral antifungal treatment.
* Individuals willing to participate in the research after receiving a full explanation of the research details, able to comply with the research procedures, and have signed the informed consent form.

Exclusion Criteria:

* Presence of nail abnormalities caused by other diseases or conditions.
* Pregnant or breastfeeding.
* History of receiving oral antifungal agents within the past 6 months or topical antifungal agents within the past 1 month prior to enrollment.
* History of photosensitivity or photodermatitis.
* Known allergy to methylene blue.
* Presence of erythematous or oedematous inflammatory skin conditions near the site of onychomycosis.
* Severe peripheral arterial disease.
* Uncontrolled diabetes mellitus or HbA1C > 8%.
* Immunocompromised status, such as HIV infection with CD4 count < 200 cells/mm³ or diagnosis of Acquired Immunodeficiency Syndrome (AIDS).
* Current use of immunosuppressive medications, including Tacrolimus, Azathioprine, Cyclosporine, Mycophenolate mofetil, or Prednisolone >10 mg/day.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the optimal light energy dose and treatment frequency for home-based photodynamic therapy (hPDT) for onychomycosis, using the L-Home PhoD device in combination with the KCMH Methylene Blue-Home Nail Kit. Efficacy will be assessed by mycologic | 12 weeks

SECONDARY OUTCOMES:
To evaluate the optimal light energy dose and treatment frequency for home-based photodynamic therapy (hPDT) for the treatment of onychomycosis. Efficacy will be assessed by changes in the dermoscopic Onychomycosis Severity Index (d-OSI) | 12 weeks
To evaluate the feasibility of home-based photodynamic therapy (hPDT) for the treatment of onychomycosis using the L-Home PhoD device in combination with the KCMH Methylene Blue-Home Nail Kit | 12 weeks
To assess the safety of home-based photodynamic therapy (hPDT) for the treatment of onychomycosis using the L-Home PhoD device in combination with the KCMH Methylene Blue-Home Nail Kit. | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No